CLINICAL TRIAL: NCT03334461
Title: Immunological and Regenerative Implications of Corrosion of Dental Materials in Children and Adolescents
Brief Title: Immunological and Regenerative Implications of Corrosion of Dental Materials
Acronym: IMUNODENT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rijeka (Other)
Collaborators: Croatian Science Foundation (Other Government)
Responsible Party: Principal Investigator, Stjepan Spalj, Full Professor, University of Rijeka
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IP-2014-09-7500
Record Dates: First submitted 2017-10-30; First posted 2017-11-07 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Caries; Enamel; Gingivitis
Keywords: Oral antiseptics; remineralisation agents
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Intervention Model Description: Randomized controlled trail
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Unlabeled bottles containing testing agent

ARMS (3):
- high concentration enamel remineralisation agent (Experimental): first month brushing teeth three times per day: twice per day with high-fluorides gel (Mirafluor K gel cola 6150 ppm F pH 5.1) and once per day without toothpaste and fluoride gel next two months brushing teeth three times per day with toothpaste containing low concentration of fluorides (1450 ppm)
  Interventions: Combination Product: Exposure to oral antiseptics or enamel remineralisation agent
- oral antiseptic (Experimental): first month brushing teeth without toothpaste three times per day and using oral antiseptic chlorhexidine mouthwash (Curasept ADS 212 a 200ml 0,12%) twice per day next two months brushing teeth three times per day with toothpaste containing low concentration of fluorides (1450 ppm)
  Interventions: Combination Product: Exposure to oral antiseptics or enamel remineralisation agent
- Control (No Intervention): regular oral hygiene without exposure to oral antiseptic or high concentration enamel remineralisation agent three months brushing teeth three times per day with toothpaste containing low concentration of fluorides (1450 ppm)

INTERVENTIONS:
Combination Product: Exposure to oral antiseptics or enamel remineralisation agent
  Arms: high concentration enamel remineralisation agent; oral antiseptic

SUMMARY:
During orthodontic treatment intraoral corrosion results with release of nickel and titanium ions from orthodontic appliances in surrounding tissues. Those transported in the saliva and blood may cause a series of side effects from hypersensitivity reactions and soft tissue proliferation to cyto and genotoxicity. Nickel is one of the strongest contact allergens, present in numerous dental alloys. The aim of this project is to investigate the immune potential of nickel and titan ions (development of allergies, changes in cariogenic potential of dental plaque, resistance of gingivitis to therapy, and bacterial resistance to antibiotics) and changes in performance of orthodontic appliances with repercussion on regeneration of bone and periodontal tissues.

DETAILED DESCRIPTION:
Tooth movement with appliances based on nickel and titanium has got great osteogenic potential and can regenerate deficient parts of alveolar bone and gingiva and rehabilitate compromised occlusal relations and a patient's masticatory function. Due to the extended duration of this therapy, different procedures are carried out and materials are applied for prevention and regeneration of damaged enamel and oral mucosa. The oral cavity may be considered a galvanic cell in which dental alloys act as electrodes, while saliva and oral preventive and regenerative agents act as electrolites. The interaction causes corrosion, reduction of elasticity and increase of stiffness of appliances, which may in turn result in excessive forces, a disruption of tissue regeneration and irreparable damage of tooth roots, surrounding alveolar bone, periodontal ligament, gingiva and pulp.

During the extended exposion, released corrosive products in surrounding tissues and those transported in saliva and blood may cause a series of side effects from hypersensitivity reactions and soft tissue proliferation to cyto and genotoxicity. Today, allergies are ever more frequent and arise earlier in life. A specific group are children and young adolescents in pubertal growth, a period in which the immune system develops. Nickel is one of the strongest contact allergens, present in numerous dental alloys. Nickel allergy is occurs in up to 28.5% of population and cannot be deemed as low potential risk anymore.

In contrast, titan was considered a biocompatible material of no allergic potential. However, there is an increase in the frequency of presentations of different hypersensitivity reactions to titan, especially in patients with pacemakers. Numerous patients with hip endoprostheses, stents, dental implans and orthodontic appliances are exposed to titan. Titan allergy may be the cause of unexplained cases of failure and rejection of dental implants. Nickel and titan could cause bacterial resistance to antibiotics which may complicate treatment of a series of infections that are more frequent in children and adolescents.

Regulations for safety of medical products regulate safety issues of materials through mandatory laboratory testing and expertise. However, the testing of interactions of these materials with newly formed materials for prevention of damage and regeneration of orodental tissues is not obligatory prior to the start of their commercial use. Such testing should be conducted by independent scientific insitutions and not by producers with direct commercial interest.

The aim of this project is to investigate:

1. the corrosion of dental materials and appliances based on nickel and titan (in saliva and due to interaction with probiotics, remineralising agents and antiseptics)
2. the immune potential of nickel and titan ions (development of allergies, changes in cariogenic potential of dental plaque, resistency of gingivitis to therapy, and bacterial resistance to antibiotics)
3. the effect of nickel and titan ions cellular level
4. changes in performance of dental appliances with repercussion on regeneration of bone and periodontal tissues.

ELIGIBILITY:
Inclusion Criteria:

* patients with fixed orthodontic appliances
* must be able to do a mouthwash

Exclusion Criteria:

* patients allergic to fluoride agents and chlorhexidine gluconate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
Reaction of oral bacterial flora to oral antiseptics and dental remineralisation agents | 30 days
  Detection of change of count of Streptococcus mutans, sorbinus and salivarius and total bacterial count assesed by qPCR in the dental plaque before and after intervention in patients with fixed orthodontic appliances.

SECONDARY OUTCOMES:
Dental arch shape | 90 days
  Measuring anterior and posterior dental arch width (in millimeters), anterior depth and depth to width ratio in orthodontic patients wearing uncoated nickel-titanium 0.020''x0.020'' archwire on the day of putting the archwire and on the day of removing it.
Oral hygiene | 210 days
  Assessing accumulation of dental biofilm with Modified Silness and Loe Plaque Index (0-3; 0=no plaque and 3=continuous line of dental bacterial plaque more than 1 millimetre).
pH of dental biofilm | 210 days
  Measuring pH of dental biofilm (colorimetric test with pH scale range from 4 to 7).
Gingivitis | 210 days
  Assessing extent of gingivitis by Full Mouth Bleeding Score (percentage).
Corrosion of dental alloy | 90 days
  Potential of corrosion, passive film breakdown and repassivation (mV)
Surface roughness of dental alloy | 90 days
  Surface roughness assessed by Atomic Force Microscopy (nm)
Friction of dental alloy | 90 days
  Friction coefficient (no units)
Forces produced by dental alloy | 90 days
  Load and unload forces measured by three-point bend test (N)
Hardness of dental alloy | 90 days
  Vickers Pyramid Number (HV)
Stifness of dental alloy | 90 days
  Young's modulus and yield strength (GPa)
Elasticity of dental alloy | 90 days
  Modulus of resilience and springback ratio (MJ/m-3)

CONTACTS AND LOCATIONS:
Overall Officials: Stjepan Spalj, PhD, Principal Investigator — University of medicine Rijeka
Locations (1):
- University of Rijeka Faculty of Dental Medicine, Rijeka, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Belasic TZ, Pejova B, Curkovic HO, Kamenar E, Cetenovic B, Spalj S. Influence of intraoral application of antiseptics and fluorides during orthodontic treatment on corrosion and mechanical characteristics of nickel-titanium alloy in orthodontic appliances. Angle Orthod. 2021 Jul 1;91(4):528-537. doi: 10.2319/052620-480.1. PMID 33566077
- [Result] Zibar Belasic T, Zigante M, Perkovic V, Uhac M, Spalj S. Comparison of dental and periodontal condition of patients unexposed and exposed to metal orthodontic appliance. Book of Abstracts of the 7th international Congress of School of Dental Medicine University of Zagreb, Rovinj, Croatia, 21.-22.05.2021. Acta Stomatol Croat. 2021;55:213-6.
- [Result] Zibar Belasic T, Zigante M, Uhac M, Karlovic S, Jelovica Badovinac I, Spalj S. Influence of intraoral application of antiseptics and fluorides during orthodontic treatment on biomechanics of remodeling of dental arches. 8th Virtual World Congress of Dental Students - Abstract book. Zagreb, Croatia, 2020. p. 2.
- [Result] Cindric L, Mohar Vitezić B, Zigante M, Spalj S, Markova Car E. Changes of bacterial profile of dental biofilm during orthodontic treatment and influence of fluorides and chlorhexidine. South Eur J Orthod Dentofac Res. Conference proceedings - 1st Congress of the Faculty of Dental medicine, University of Rijeka, Croatia, October 1st-3rd 2020. Rijeka, Hrvatska, 2020. p. 55.
- [Result] Zibar Belasic T, Pejova B, Otmacic Curkovic H, Kamenar E, Cetenovic B, Spalj S. Intraoral application of antiseptics and fluorides during orthodontic treatment does not affect significantly corrosion and mechanical characteristics of nickel-titanium alloy in orthodontic appliances. Prvi kongres Fakulteta dentalne medicine Sveučilišta u Rijeci, Rijeka, 1-2.10.2020. Knjiga sažetaka. South Eur J Orthod Dentofac Res 2020;7:56.
- [Result] Zibar Belasic T, Mohar Vitezic B, Zigante M, Spalj S, Markova Car E. Supragingival biofilm composition changes during orthodontic treatment and chlorhexidine use. Book of Abstracts 97th Annual Congress of the European Orthodontic Society, Limassol, Cipar, 30.05.-03.06.2022.
- See also: all data concerning research project are available at link (Immune and regenerative implications of corrosion of dental materials in children and adolescents) — http://arhiva.medri.uniri.hr/~spaljs/
- See also: all data concerning new project are available at link (Environmental factors and microbiological interactions in the structure of dental biofilm) — https://sites.google.com/view/ip-2020-02/početna-stranica